CLINICAL TRIAL: NCT05176795
Title: Study of the Determinants of Pediatric Onset Inflammatory Diseases: Host-microbiota-environment Interactions
Brief Title: Host-microbiota-environment Interactions
Acronym: MIP-1
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 MERLIN; 2021-AO1006-35 (Other: ANSM)
Record Dates: First submitted 2021-12-14; First posted 2022-01-04 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2021-12

CONDITIONS: Juvenile Idiopathic Arthritis; Diabetes type1; Inflammatory Bowel Diseases
Keywords: microbiota; environmental factors; food contaminants
MeSH Terms: conditions — Arthritis, Juvenile; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: Child under 10 years old newly diagnosed with JIA, IBD or T1DM
  Interventions: Other: Stool sample
- Active Comparator: Healthy control: Brother/sister of child with pediatric onset inflammatory disease (same age category - same environment: food, living space)
  Interventions: Other: Stool sample

INTERVENTIONS:
Other: Stool sample — Comparaison of the gut microbiota composition

SUMMARY:
Two types of inflammatory and autoimmune diseases (excluding monogenic diseases) can be distinguished in children: those similar to adult diseases but with an early onset (type 1 diabetes, inflammatory diseases of the gastrointestinal tract, rheumatoid arthritis with anti-CCP antibodies) and those specific to children that are not described in adults (early-onset juvenile idiopathic arthritis with anti-nuclear and anterior uveitis).

The familial and nosological aggregations suggest that these diseases are probably polygenically determined, and result from interactions with the environment. In a singular way, the incidence of "adult" diseases is increasing while the age of onset is getting earlier; conversely, there is no increase in early-onset juvenile idiopathic arthritis.

On the other hand, the influence of early events that may alter the microbiotic environment is different for different diseases: whereas cesarean section (or early antibiotic therapy) has been shown to increase the risk of JIA and T1DM, it does not seem to change the risk of IBD. We hypothesize that environmental factors, particularly those related to diet and bacterial and fungal digestive microbiota - are different between these disease categories.

DETAILED DESCRIPTION:
Exploratory pathophysiology monocentric study including an initial case-control study, followed by a cohort for cases.

Controls will be siblings of cases with longitudinal follow-up.

Stool samples will be collected simultaneously from the child with JIA, T1DM or IBD (case) and his/her sibling(s) (control):

* at the time of diagnosis
* two months after diagnosis (for children with inflammatory disease only)
* one year after diagnosis (cases and controls)

Tryptase level in plasma will be recorded for the child with JIA, T1DM or IBD (at the time of diagnosis, 2 months and 1 year after diagnosis)

ELIGIBILITY:
Inclusion Criteria:

CASE:

- Newly diagnosed with JIA, IBD or T1DM

CONTROL:

- Brother/sister of child with pediatric onset inflammatory disease (same age category - same environment: diet, living environment)

Exclusion Criteria (case and control):

* Child with antibiotic treatment in the 4 weeks preceding the stool sample
* Recent digestive infectious disease (bacterial, viral, parasitic) (end of episode < 7 days)

Exclusion Criteria (control): children with autoimmune or inflammatory disease

Ages: 0 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The participants include patient-sibling pairs meeting the inclusion criteria (30 children newly diagnosed with JIA, IBD or T1DM and 30 siblings).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota composition | Day 1
  Variation between cases and controls in gut microbiota composition (determination of the gut microbiota composition by 16S metagenomic)
Gut microbiota composition | 12 months
  Variation between cases and controls in gut microbiota composition (determination of the gut microbiota composition by 16S metagenomic)

SECONDARY OUTCOMES:
Composition of the fecal volatolome | Day 1
  The volatile compounds in the samples will be analyzed via solid-phase microextraction (SPME) coupled with gas chromatography-mass spectrometry (GC-MS)
Variation in gut microbiota following initiation of therapy in patients newly diagnosed with JIA, IBD or T1DM. | Day 1, 2 months, 12 months
  Characterization of the gut microbiota using a capture method by hybridization of the gene encoding 16S rRNA
Tryptasemia | Day 1, 2 months, 12 months
  Variation in plasma tryptase levels during the first year of the disease
Fecal contamination with nanoparticles | Day 1
  measurement of titane and silicia levels in stool sample

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Merlin, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwiertz A, Jacobi M, Frick JS, Richter M, Rusch K, Kohler H. Microbiota in pediatric inflammatory bowel disease. J Pediatr. 2010 Aug;157(2):240-244.e1. doi: 10.1016/j.jpeds.2010.02.046. Epub 2010 Apr 18. PMID 20400104
- [Background] Rouxel O, Da Silva J, Beaudoin L, Nel I, Tard C, Cagninacci L, Kiaf B, Oshima M, Diedisheim M, Salou M, Corbett A, Rossjohn J, McCluskey J, Scharfmann R, Battaglia M, Polak M, Lantz O, Beltrand J, Lehuen A. Cytotoxic and regulatory roles of mucosal-associated invariant T cells in type 1 diabetes. Nat Immunol. 2017 Dec;18(12):1321-1331. doi: 10.1038/ni.3854. Epub 2017 Oct 9. PMID 28991267
- [Background] Di Paola M, Cavalieri D, Albanese D, Sordo M, Pindo M, Donati C, Pagnini I, Giani T, Simonini G, Paladini A, Lionetti P, De Filippo C, Cimaz R. Alteration of Fecal Microbiota Profiles in Juvenile Idiopathic Arthritis. Associations with HLA-B27 Allele and Disease Status. Front Microbiol. 2016 Oct 26;7:1703. doi: 10.3389/fmicb.2016.01703. eCollection 2016. PMID 27833598
- [Background] Defois C, Ratel J, Garrait G, Denis S, Le Goff O, Talvas J, Mosoni P, Engel E, Peyret P. Food Chemicals Disrupt Human Gut Microbiota Activity And Impact Intestinal Homeostasis As Revealed By In Vitro Systems. Sci Rep. 2018 Jul 20;8(1):11006. doi: 10.1038/s41598-018-29376-9. PMID 30030472